CLINICAL TRIAL: NCT00883259
Title: Metformin Treatment for Preventing Gestational Diabetes in High-risk Patients
Brief Title: Metformin and Gestational Diabetes in High-risk Patients: a RCTs
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Stefano Palomba, Associate Professor, University Magna Graecia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 12/2008
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Obesity; Polycystic Ovary Syndrome; Gestational Diabetes
Keywords: High-risk patients; Metformin; PCOS; Pregnancy complications; Previous gestational DM
MeSH Terms: conditions — Obesity; Polycystic Ovary Syndrome; Diabetes, Gestational; Pregnancy Complications | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): Metformin treatment
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Placebo tablets
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Metformin — 850 mg twice daily
  Arms: Experimental
Other: Placebo — Microcristallyne cellulose 1 table twice daily
  Arms: Placebo

SUMMARY:
Gestational diabetes mellitus (DM) is one of the most frequent complications in pregnant patients with polycystic ovary syndrome (PCOS) in 20-40% of cases and ~40% of patients with gestational DM are likely to have underlying polycystic ovarian morphology. A recent meta-analysis demonstrated a significantly higher risk of developing gestational DM [odds ratio (OR) 2.94; 95% confidence interval (CI): 1.70-5.08] in the PCOS population.

Metformin is an oral biguanide insulin sensitizer used for treating type-2 DM and recently introduced to treat PCOS.

At the moment, preliminary data seem to reassure regarding the use of metformin in PCOS patients showing benefits for maternal and fetal outcomes, without serious adverse events. Furthermore, well-designed randomized, controlled trials (RCTs) on this issue are lacking, thus it is not possible to either suggest or advice against the use of metformin during pregnancy for reducing gestational DM risk. To this regard, PCOS represents an intriguing model of "high-risk patients" to evaluate the efficacy of metformin for preventing DM development.

The present protocol firstly will evaluate the effects of metformin administration in reducing incidence of gestational DM in high-risk patients, such as pregnant PCOS patients.

DETAILED DESCRIPTION:
Obese pregnant PCOS patients with previous diagnosis of gestational DM will be enrolled and allocated into two treatment arms (experimental and placebo groups). Subjects in the experimental group will receive metformin at dosage of 850 mg twice daily, whereas subjects in the control group will receive placebo tablets (microcristallyne cellulose) twice daily.

At baseline, all subjects will undergo clinical evaluation, serial ultrasound examinations, and venous blood drawing to evaluate complete hormonal assays and serum fasting glucose and insulin levels. The homeostasis model of assessment-insulin resistance, the fasting glucose-to-insulin ratio, and the free androgen index will be also calculated. Monthly follow-up visits will be performed for assessing maternal and fetal wellbeing.

The primary endpoint of the study will be the incidence of gestational DM. The power analysis and the sample size calculation, performed using SamplePower release 2.0, showed that we will need to enroll at least 40 patients for each group to yield a statistically significant result with a power study of 90%. For categorical variables, the Pearson chi-square test will be performed. Continuous data will be expressed either as mean and standard deviation or median and inter-quartile range with min-max values, according to their normal distribution, and analysed using the Student t test or Mann-Whitney U test, respectively. Statistical significance will be set at P<0.05. The Statistics Package for Social Science (SPSS 14.0.1; Chicago, IL, USA) will be used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with Polycystic Ovary Syndrome (using ASRM/ESHRE criteria)
* BMI > 30
* Previous diagnosis of gestational DM

Exclusion Criteria:

* Major medical conditions
* Organic pelvic diseases
* Previous pelvic surgery

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-09; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of gestational DM in high-risk patients | 36 months

SECONDARY OUTCOMES:
Abortion | 36 months
Pregnancy-induced hypertension | 36 months
Pre-eclampsia | 36 months
Macrosomia | 36 months
Fetal malformations | 36 months
Premature deliveries | 36 months
Intrauterine deaths | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Palomba, MD, Principal Investigator — Department of Obstetrics & Gynecology - University Magna Graecia of Catanzaro; Francesco Orio, MD, Principal Investigator — Endocrinology - University " Parthenope" of Naples; Achille Tolino, MD, Principal Investigator — Department of Obstetrics & Gynecology, University of Naples; Tommaso Simoncini, MD, Principal Investigator — Department of Obstetrics & Gynecology - University of Pisa; Fulvio Zullo, MD, Principal Investigator — Gynecologic Unit, Cancer Center of Excellence "Tommaso Campanella" of Catanzaro
Locations (3):
- Italy (3):
  - Pugliese Hospital, Catanzaro, Catanzaro, CZ
  - "Pugliese" Hospital, Catanzaro, Catanzaro
  - University of Catanzaro, Italy, Catanzaro